CLINICAL TRIAL: NCT05453357
Title: Feasibility and Acceptability of a Remote Glucose Monitoring Program for Pregnant Marshallese Women with Pregnancies Complicated by Diabetes
Brief Title: Feasibility and Acceptability of a Remote Glucose Monitoring Program for Pregnant Marshallese Women
Status: Withdrawn | Type: Observational
Why Stopped: Funding ended before enrollment
Sponsor: University of Arkansas (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 274147; UL1TR003107 (NIH); KL2TR003108 (NIH)
Record Dates: First submitted 2022-07-06; First posted 2022-07-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-04

CONDITIONS: Diabetes, Gestational; Diabetes Mellitus Type 2 Pre-Existing
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- iGlucose Remote Glucose Monitoring: Patients will be provided with the iGlucose monitor at baseline data collection.
  Interventions: Device: iGlucose

INTERVENTIONS:
Device: iGlucose — The patient will use the monitor as instructed by their healthcare team to monitor their blood glucose.

SUMMARY:
The overall objective is to test the feasibility and acceptability of a remote glucose monitoring program among Marshallese women with PGDM (pre-gestational diabetes mellitus) or GDM (gestational diabetes mellitus) and with limited English proficiency.

DETAILED DESCRIPTION:
iGlucose Remote Monitoring System. iGlucose is a remote patient monitoring system. The iGlucose monitor works by analyzing a small amount of blood placed on a strip that is inserted into the monitor, similar to a standard glucometer. The iGlucose monitor will show the patient their glucose reading and will automatically send the patient's glucose reading to a database via cellular networks when the patient removes the strip from the device. The iGlucose monitor does not require any recording on the part of the patient. The iGlucose data is managed through a HIPAA-compliant Amazon Web Services (AWS) database maintained by Smartmeter. The data is available to the provider to monitor the patient's blood glucose levels accurately and in a timely manner, allowing for treatment to be adjusted. The data is available for the physician during every patient contact for review and discussion.

Patients will be provided with the iGlucose monitor at the baseline data collection. A trained bilingual research assistant will review the iGlucose guide with the participant, provide training on the use of the monitor, taking a blood glucose reading with the monitor, and the patient will use the iGlucose monitor once in front of the research assistant. The patient will receive a packet of information in their language of choice (English and/or Marshallese). The packet will include information on how to use the monitor (including the iGlucose Guide) and contact information if there are any problems with the monitor during the study. The patient will use the monitor as instructed by their healthcare team to monitor their blood glucose. The patient will return the equipment at the completion of the study.

The participant will provide their physician's information as part of the study, so that the investigators may provide access to the iGlucose blood glucose readings through the electronic guidebook and contact the physician post-intervention to complete a survey.

ELIGIBILITY:
Inclusion Criteria:

* Women who self-identify as Marshallese
* 18 years of age or older
* ≤30 weeks pregnant
* Receive prenatal care at University of Arkansas for Medical Sciences (UAMS) and partner clinics and hospitals
* Have used a paper log for at least two weeks
* Have a diagnosis of PGDM (pre-gestational diabetes mellitus) or GDM (gestational diabetes mellitus).

Exclusion Criteria:

* Women who are unable to use a glucometer by themselves
* Have not used a paper log
* Have a continuous glucose monitor
* More than 30 weeks pregnant

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Twenty Marshallese women with pregestational or gestational diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Overall Acceptability of Remote Glucose Monitoring | Change in baseline glucose monitoring satisfaction score at two weeks postpartum
  The investigator will conduct a t-test (α=.05) using the post-intervention scores on the glucose monitoring satisfaction survey given to participants; a higher mean score demonstrating more satisfaction with the iGlucose remote monitoring system (range 0-60). The semi-structured interview qualitative data will be analyzed to explore the feasibility and acceptability of the intervention qualitatively. The investigator will use descriptive statistics to assess physician satisfaction with the iGlucose remote monitoring system. Given the small size of the pilot study, the investigator will conduct a review of the disaggregated data to determine the individual differences between pre- and post-intervention scores on the glucose monitoring satisfaction measure to better understand the changes in glucose monitoring satisfaction.
Overall Feasibility of Remote Glucose Monitoring | Retention at two weeks postpartum
  The investigator will use summary statistics to document and compare actual recruitment and retention rates with the target rates. A recruitment rate of ≥70% of all eligible participants, a retention rate through postnatal data collection of ≥80%, and an engagement rate of ≥75% of recommended daily glucose checks completed during the enrollment period will indicate feasibility.

SECONDARY OUTCOMES:
Changes in patient-physician communication | Change in baseline Assessment of Care for Chronic Conditions+ (ACC+) score at two weeks postpartum
  The investigator will conduct repeated measures t-test (α=.05) using pre- and post-intervention patient satisfaction with patient-physician communication scores from the Assessment of Care for Chronic Conditions+ (ACC+) survey measures. The repeated measures t-test will assess whether the post-intervention mean ACC+ score (range 0-100) is significantly higher than the pre-intervention score, indicating increased patient satisfaction with patient-physician communication.
Changes in self-efficacy | Change in baseline self-efficacy score at two weeks postpartum
  The investigator will conduct repeated measures t-test (α=.05) using pre- and post-intervention self-efficacy scores from the Diabetes Management Self-Efficacy Scale (DMSES) (range 0-80).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Andersen, PhD, Principal Investigator — University of Arkansas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McElfish PA, Rowland B, Long CR, Hudson J, Piel M, Buron B, Riklon S, Bing WI, Warmack TS. Diabetes and Hypertension in Marshallese Adults: Results from Faith-Based Health Screenings. J Racial Ethn Health Disparities. 2017 Dec;4(6):1042-1050. doi: 10.1007/s40615-016-0308-y. Epub 2016 Nov 11. PMID 27837454
- [Background] Bogdanet D, Egan A, Reddin C, Kirwan B, Carmody L, Dunne F. ATLANTIC DIP: Despite insulin therapy in women with IADPSG diagnosed GDM, desired pregnancy outcomes are still not achieved. What are we missing? Diabetes Res Clin Pract. 2018 Feb;136:116-123. doi: 10.1016/j.diabres.2017.12.003. Epub 2017 Dec 15. PMID 29253626
- [Background] Alexopoulos AS, Blair R, Peters AL. Management of Preexisting Diabetes in Pregnancy: A Review. JAMA. 2019 May 14;321(18):1811-1819. doi: 10.1001/jama.2019.4981. PMID 31087027
- [Background] Sushko K, Menezes HT, Strachan P, Butt M, Sherifali D. Self-management education among women with pre-existing diabetes in pregnancy: A scoping review. Int J Nurs Stud. 2021 May;117:103883. doi: 10.1016/j.ijnurstu.2021.103883. Epub 2021 Jan 20. PMID 33548591
- [Background] American Diabetes Association. 14. Management of Diabetes in Pregnancy: Standards of Medical Care in Diabetes-2020. Diabetes Care. 2020 Jan;43(Suppl 1):S183-S192. doi: 10.2337/dc20-S014. PMID 31862757
- [Background] Berger H, Gagnon R, Sermer M, Basso M, Bos H, Brown RN, Bujold E, Cooper SL, Gagnon R, Gouin K, McLeod NL, Menticoglou SM, Mundle WR, Roggensack A, Sanderson FL, Walsh JD. Diabetes in Pregnancy. J Obstet Gynaecol Can. 2016 Jul;38(7):667-679.e1. doi: 10.1016/j.jogc.2016.04.002. Epub 2016 May 12. PMID 27591352
- [Background] Schaefer-Graf U, Napoli A, Nolan CJ; Diabetic Pregnancy Study Group. Diabetes in pregnancy: a new decade of challenges ahead. Diabetologia. 2018 May;61(5):1012-1021. doi: 10.1007/s00125-018-4545-y. Epub 2018 Jan 22. PMID 29356835
- [Background] Goyal S, Cafazzo JA. Mobile phone health apps for diabetes management: current evidence and future developments. QJM. 2013 Dec;106(12):1067-9. doi: 10.1093/qjmed/hct203. Epub 2013 Oct 8. PMID 24106313
- [Background] Guo H, Zhang Y, Li P, Zhou P, Chen LM, Li SY. Evaluating the effects of mobile health intervention on weight management, glycemic control and pregnancy outcomes in patients with gestational diabetes mellitus. J Endocrinol Invest. 2019 Jun;42(6):709-714. doi: 10.1007/s40618-018-0975-0. Epub 2018 Nov 7. PMID 30406378
- [Background] Andersen JA, Scoggins D, Michaud T, Wan N, Wen M, Su D. Racial Disparities in Diabetes Management Outcomes: Evidence from a Remote Patient Monitoring Program for Type 2 Diabetic Patients. Telemed J E Health. 2021 Jan;27(1):55-61. doi: 10.1089/tmj.2019.0280. Epub 2020 Apr 17. PMID 32302521
- [Background] Mora P, Buskirk A, Lyden M, Parkin CG, Borsa L, Petersen B. Use of a Novel, Remotely Connected Diabetes Management System Is Associated with Increased Treatment Satisfaction, Reduced Diabetes Distress, and Improved Glycemic Control in Individuals with Insulin-Treated Diabetes: First Results from the Personal Diabetes Management Study. Diabetes Technol Ther. 2017 Dec;19(12):715-722. doi: 10.1089/dia.2017.0206. Epub 2017 Oct 13. PMID 29027812
- [Background] Diamond L, Izquierdo K, Canfield D, Matsoukas K, Gany F. A Systematic Review of the Impact of Patient-Physician Non-English Language Concordance on Quality of Care and Outcomes. J Gen Intern Med. 2019 Aug;34(8):1591-1606. doi: 10.1007/s11606-019-04847-5. Epub 2019 May 30. PMID 31147980